CLINICAL TRIAL: NCT00901680
Title: Creation of the BioBank,To Establish a Multidisciplinary Research Structure That Facilitates Projects That Bridge Specialties That Normally May or May Not Interact.
Brief Title: Creation of the BioBank, Early Detection and Discovery Biomarkers
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, George Wilson, George Wilson PhD, Corewell Health East
Other Study IDs: HIC 2008-180
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Pancreatic Cancer; Head and Neck Cancer; Breast Cancer
Keywords: Tissue Bank
MeSH Terms: conditions — Pancreatic Neoplasms; Head and Neck Neoplasms; Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens to be retained are tissue, blood, whole blood, DNA, RNA, urine saliva,cerebral spinal fluid, amniotic fluid.
Oversight: Data Monitoring Committee: No

SUMMARY:
To establish a multidisciplinary research structure for tissue repository that facilitates projects that bridge specialties that normally may or may not interact.

DETAILED DESCRIPTION:
To establish a multidisciplinary research structure that facilitates projects that bridge specialties that normally may or may not interact. The tissue bank will build the platform for a novel application of translational research that links cutting edge molecular laboratory techniques to clinical outcome studies in a fast and direct manner. Tissue banks can be used for numerous discovery applications such as the identification and structural characterization of human genes, expression analysis, or discovery proteomics. Biological specimens, when coupled with standardized treatment and outcome data, will be essential resources for the identification, characterization, and validation of biomarkers that are predictive of disease and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers

Exclusion Criteria:

* N/A volunteers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population male/female from inpatient and outpatient hospital settings or doctor offices..
Sampling Method: Non-Probability Sample
Enrollment: 3028 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wilson, PhD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospitals, Royal Oak, Michigan, United States